CLINICAL TRIAL: NCT05189327
Title: Non-interventional Observational Prospective Longitudinal Study of the Incidence of Ulcerative Colitis and Crohn's Disease Among the Adult Population of the Republic of Kazakhstan
Brief Title: Noninterventional Observational Prospective Longitudinal Study of the Incidence of Ulcerative Colitis and Crohn's Disease Among the Adult Population of the Republic of Kazakhstan
Acronym: NUCaCD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Kazakhstan Scientific Society for Study of intestine diseases (Other)
Collaborators: FERRING Kazakhstan (Unknown)
Responsible Party: Sponsor
Other Study IDs: KSSSID-052021
Record Dates: First submitted 2021-12-29; First posted 2022-01-12 (Actual); Last update posted 2022-01-12 (Actual); Status verified 2021-12

CONDITIONS: Ulcerative Colitis Chronic; Crohn Disease Colon
Keywords: Nonspecific Ulcerative colitis; Crohn Disease; Patient Registry
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with diagnosed Nonspecific Ulcerative Colitis and Crohn Disease: All patients with diagnosed Nonspecific Ulcerative Colitis and Crohn Disease in the Republic of Kazakhstan.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — Non-interventional study

SUMMARY:
The NUCaCD study aims to develop a reliable registry of patients suffering inflammatory bowel diseases in the Republic of Kazakhstan.

DETAILED DESCRIPTION:
The NUCaCD aims to study the prevalence of inflammatory bowel diseases in the Republic of Kazakhstan and create a reliable database, which will greatly facilitate future planning of the volume of health resources needed to address these diseases management and will help to optimize preventive measures and will support future research to better understand the etiology, new options treatment and factors affecting prognosis, relapses, development of complications and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Availability of a signed informed consent form; or the presence of a disinterested witness if the patient is unable to examine and sign the consent form due to illiteracy or disability (for example, in the case of blindness);
* The patient has a documented diagnosis of ulcerative colitis or Crohn's disease (endoscopy, histology, if indicated by radiation diagnostics);
* Patients who have applied for treatment or are already taking treatment from a gastroenterologist / coloproctologist, including inpatients;
* Citizenship of the Republic of Kazakhstan (or resides).

Exclusion Criteria:

* Patient takes part in an interventional clinical trial;
* Patient is unable to follow the schedule of the visits;
* Any condition that the PI believes would prevent a study participant from participating in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with a verified diagnosis of Nonspecific Ulcerative Colitis and Crohn Disease.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2021-12-10 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
To study the incidence of NUC and CD in the Republic of Kazakhstan | 2 years
  To study the incidence of NUC and CD in the Republic of Kazakhstan

SECONDARY OUTCOMES:
To study the patterns of the course of the disease and the treatment effect | 2 years
  To study the patterns of the course of the disease and the effectiveness of drug therapy in outpatient and inpatient clinics.
Conduct an analysis of the completeness of the diagnosis and compliance with the national guidelines for the diagnosis and treatment of ulcerative colitis and Crohn's disease | 2 years
  Conduct an analysis of the completeness of the diagnosis and compliance with the national guidelines for the diagnosis and treatment of ulcerative colitis and Crohn's disease
Analysis of the relationship between management strategies and treatment outcomes | 2 years
  Analysis of the relationship between management strategies and treatment outcomes

CONTACTS AND LOCATIONS:
Overall Officials: Jamilya Kaibullayeva, PhD, Study Director — KSSSID
Locations (1):
- Primary Health Clinic #5, Almaty, Kazakhstan

IPD SHARING:
Plan to Share IPD: No